CLINICAL TRIAL: NCT03045536
Title: Evaluation of Partial and Total Femoral Replacement Treated in a Single Orthopedic Centre
Brief Title: Evaluation of Partial and Total Femoral Replacement
Acronym: EFeRe
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Technical University of Munich (Other)
Responsible Party: Principal Investigator, Harrasser, Principal Investigator, Technical University of Munich
Other Study IDs: 148/15
Record Dates: First submitted 2017-02-04; First posted 2017-02-07 (Estimated); Last update posted 2017-04-25 (Actual); Status verified 2017-02

CONDITIONS: Survival, Prostheses

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with TFR: Patients treated with TFR for oncologic or non-oncologic reason
  Interventions: Device: MML (Fa. ESKA/Orthodynamics)

INTERVENTIONS:
Device: MML (Fa. ESKA/Orthodynamics) — Classification of complications according to MSTS

SUMMARY:
Several surgical options for the reconstruction of massive bone defects have been described and include biologic methods with autografts and allografts, and the use of tumor endoprostheses (total femoral replacement, TFR). Several types of modular TFR are available, but nevertheless unpredictable outcomes and high complication rates have been described from most authors. The aim of the present study was to compare complication rates after TFR performed with modular total femur prosthesis MML (Fa. ESKA/Orthodynamics) in patients with and without malignant disease.

ELIGIBILITY:
Inclusion Criteria:

* Total or partial femoral replacement

Exclusion Criteria:

* Failure of device

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The investigators retrospectivel review our institution's database for patients who underwent resection of the partial or whole femur due to bone tumors or failed revision arthroplasties and reconstruction by TFR from January 1995 to January 2011.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2016-01-01 (Actual); Primary Completion 2018-03-01 (Estimated); Study Completion 2019-04-01 (Estimated)

PRIMARY OUTCOMES:
Survival of device | 2 years
  Any device-related complications are defined failure

CONTACTS AND LOCATIONS:
Overall Officials: norbert harrasser, Principal Investigator — Klinikum rechts der Isar
Locations (1):
- Klinikum rechts der Isar, Munich, Germany

IPD SHARING:
Plan to Share IPD: No